CLINICAL TRIAL: NCT00523198
Title: Correlation Between Salivary Cortisol and Free Serum Cortisol Compared to Total Serum Cortisol in MICU Patients With Septic Shock
Brief Title: Correlation Salivary Cortisol and Free Serum Cortisol to Total Serum Cortisol in MICU Septic Shock
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Rosa Estrada Y Martin, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-06-413; M01-RR 02558 (GCRC) (Other: Memorial Hermann Hospital); M01RR002558 (NIH)
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Septic Shock
Keywords: Cortisol
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is:

* to correlate salivary cortisol to free serum cortisol (as salivary cortisol is considered to be almost complete free cortisol) and,
* to correlate free serum cortisol to total serum cortisol levels

Both in patients with septic shock (severe sepsis requiring vasopressors).

We believe that:

* total serum cortisol does not correlate with free serum cortisol in patient with septic shock and,
* that salivary cortisol correlates with free serum cortisol and can be used to determine the level of free serum cortisol.

DETAILED DESCRIPTION:
Free serum cortisol is considered the active hormone.

In patients with septic shock only the total serum cortisol level is available, however, the free cortisol level can be normal despite a low total cortisol level due to changes in the serum protein.

The hormone can be replaced improperly in these patients and contribute to poor outcome in septic shock.

We are studying adult MICU patients with septic shock who are not receiving corticosteroid replacement.

This study does not include any intervention.

In-hospital or 28-day mortality are registered in all the patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with septic shock

Exclusion Criteria:

* Corticosteroid replacement
* Blood in mouth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MICU patients with septic shock
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-02; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Salivary cortisol | one year
  salivary cortisol in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Estrada-Y-Martin, MD, Principal Investigator — The University of Texas-Health Science Center at Houston / Division of Pulmonary, Sleep and Critical Care Medicine
Locations (1):
- The University of Texas- Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Estrada-Y-Martin RM, Orlander PR. Salivary cortisol can replace free serum cortisol measurements in patients with septic shock. Chest. 2011 Nov;140(5):1216-1222. doi: 10.1378/chest.11-0448. Epub 2011 Aug 4. PMID 21816912